CLINICAL TRIAL: NCT05739110
Title: Optimizing Hepatocellular Carcinoma Disease Staging Systems by Incorporating Tumor Micronecrosis: A Multi-institutional Retrospective Study
Brief Title: HCC Staging Modified by Tumor Micronecrosis
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Huizhou Municipal Central Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Director, Zhejiang University
Other Study IDs: HCCNSTAGE
Record Dates: First submitted 2023-02-11; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Tumor micronecrosis; BCLC; TNM; Disease staging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- micronecrosis(+) group: Hepatocellular patients with tumor micronecrosis.
  Interventions: Behavioral: tumor micronecrosis
- micronecrosis(-) group: Hepatocellular patients without tumor micronecrosis.

INTERVENTIONS:
Behavioral: tumor micronecrosis — whether HCC patients have tumor micronecrosis or not
  Groups: micronecrosis(+) group

SUMMARY:
Tumor micronecrosis is a pathological feature that reflects malignant biological behavior in hepatocellular carcinoma (HCC). This study aimed to evaluate the prognostic significance of tumor micronecrosis based on the current BCLC and TNM staging systems, and futher improve the performance of the staging models by establishing modified new staging models including tumor micronecrosis.

ELIGIBILITY:
Inclusion Criteria:

* primary and histologically confirmed HCCs
* patients who underwent curative liver resection

Exclusion Criteria:

* simultaneous presence of other tumors
* patients who had received preoperative antitumor therapies
* no available surgical specimens for evaluating micronecrosis status
* gross tumor necrosis and Nscore = 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study enrolled patients who underwent liver resection from four institutions in China: the First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU) (n = 896), Mengchao Hepatobiliary Hospital of Fujian Medical University (n = 94), the Second Affiliated Hospital of Nanchang University (n = 84), and Huzhou Central Hospital (n = 36).
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | from date after liver resection until death or last follow-up, whichever came first, assessed up to 72 months
  the number of months from the date of surgery to the date of the last follow-up visit or time of death.

SECONDARY OUTCOMES:
Disease-free survival | from date after liver resection until recurrence or last follow-up, whichever came first, assessed up to 72 months
  the number of months from the date of surgery to the date of first confirmable recurrence or death

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No